CLINICAL TRIAL: NCT01500642
Title: Comparison of the Efficacy and the Safety of Different Schedules of Administration of Sub-lingual Immunotherapy in Patients With Ragweed Pollinosis: a Phase III Randomized and Controlled Clinical Study
Brief Title: Comparison of the Efficacy and the Safety of Different Schedules of Administration of Sub-lingual Immunotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ASST Fatebenefratelli Sacco (Other)
Collaborators: ALK-Abelló A/S (Industry)
Responsible Party: Principal Investigator, Iemoli Enrico, director allergy and clinical immunology department, ASST Fatebenefratelli Sacco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130/2011/29/AP
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Pollen Allergy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- sublingual immunotherapy (Active Comparator): 15 patients treated with sublingual immunotherapy (SLIT One, ALK Abello) administered at standard dose (200 STU / dose) from June to August 2001
  Interventions: Biological: Slit One
- vestibular immunotherapy (Active Comparator): 15 patients treated with vestibular immunotherapy (SLIT One, ALK Abello) administered at standard dose (200 STU / dose) from June to August 2001
  Interventions: Biological: Slit One
- sublingual doubled immunotherapy (Active Comparator): 15 patients treated with sublingual immunotherapy (SLIT One, ALK Abello) administered at doubled dose (400 STU / dose) from June to August 2001
  Interventions: Biological: Slit One ragweed

INTERVENTIONS:
Biological: Slit One — slit one sublingual immunotherapy 200 stu
  Other Names: Slitone (Alk Abello)
  Arms: sublingual immunotherapy
Biological: Slit One — slit one vestibular immunotherapy 200 stu
  Other Names: Slitone (Alk Abello)
  Arms: vestibular immunotherapy
Biological: Slit One ragweed — slit one 400 stu dose ragweed (sublingual doubled immunotherapy)
  Other Names: Slitone (Alk Abello)
  Arms: sublingual doubled immunotherapy

SUMMARY:
The dose and the mode of administration of sublingual therapy remain open questions to determine the efficacy and safety of this desensitization therapy, the main purpose of this study is to evaluate if different routes of administration (oral-vestibular vs. sublingual) and a maximum dose of allergen administered are able to determine a different effect or a different incidence of side effects of the therapy in a group of patients with rhinoconjunctivitis and/or asthma due to ragweed

DETAILED DESCRIPTION:
Version 1 16/02/2011 The allergen-specific immunotherapy represents an important therapeutic option for the treatment of allergic respiratory diseases. Its clinical efficacy is well demonstrated, although the mechanism of action is still under study.

The main purpose of immunotherapy is to induce an allergen-specific tolerance so that the natural exposure to the allergen does not cause clinical symptoms.

The clinical efficacy of standard subcutaneous immunotherapy (SCIT) is known. A meta-analysis Cochrane on the clinical efficacy of SCIT in allergic rhinitis 51 double-blind studies with a total 2871 patients) demonstrated a reduction in symptoms in 73% of patients and a reduction in the use of drugs in 57%.

Other studies also show that SCIT was effective in the long term (at least 3-5 years of suspension) reduces sensitization to new allergens, prevents progression of allergic rhinitis in asthma and significantly improves the symptoms of asthma, hyper- bronchial reactivity and the use of asthma medications.

Sublingual immunotherapy (SLIT) represents an effective alternative route of administration of vaccine therapy with an allergic profile security than the SCIT.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-55 years
* Known allergy to ragweed pollen
* No immunotherapy or in progress prior to enrollment
* Symptoms of rhino / conjunctivitis with or without asthma

Exclusion Criteria:

* Allergic to perennial allergens (moulds, mites and animal when exposed to the animal)
* Patients with chronic diseases (infectious, autoimmune cancer, heart or kidney)
* Are pregnant
* Chronic drug treatment with steroids and / or immunosuppressive
* Oral disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the percentage of CD14-PDL-1-IL10 + circulating allergen-specific (ragweed) in pre-seasonal SLIT vs oral-vestibular regimen and in pre-seasonal regimen of SLIT at 400 STU/dose vs 200 STU | 3 months

SECONDARY OUTCOMES:
Evaluation of clinical efficacy (as assessed by symptom score and use of symptomatic drugs) among patients treated with sublingual vaccine by vestibular compared to those treated sublingually | 3 months
Evaluation of clinical efficacy (as assessed by symptom score and use of symptomatic drugs) among patients treated with sublingual vaccine dose doubled compared to those treated with standard dose | 3 months
Evaluation of the safety and tolerability (as assessed by data collection form of local and systemic adverse events) among patients treated with sublingual vaccine in oral/vestibular administration compared to those treated sublingually | 3 months
Assessment of safety and tolerability (assessed using data forms of local and systemic adverse events) among patients treated with sublingual vaccine dose doubled compared to those treated with standard dose | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: enrico iemoli, phd, Principal Investigator — luigi sacco hospital milano
Locations (1):
- Luigi Sacco Hospital, Milan, Italy